CLINICAL TRIAL: NCT02926352
Title: Effects of Low-Level Laser Stimulation With and Without Fear Extinction Training in the Modification of Pathological Fear
Brief Title: Effects of Low-Level Laser Stimulation With and Without Fear Extinction Training
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Director of the Laboratory for the Study of Anxiety Disorders, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-12-0068
Record Dates: First submitted 2015-08-28; First posted 2016-10-06 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Phobias; Claustrophobia; Social Phobia
Keywords: LLLT; LLLS; Low-Level Laser Stimulation; Low-Level Laser Therapy; Low-Level Light Therapy; Transcranial infrared light stimulation; Near-infrared light; Photobiomodulation; Fear Extinction; Exposure Therapy; Claustrophobia; Fear of enclosed spaces; Fear of contamination; Fear of public speaking; Anxiety sensitivity; Cytochrome oxidase; Memory consolidation; Cognitive enhancer
MeSH Terms: conditions — Phobic Disorders; Claustrophobia; Phobia, Social; Glossophobia | interventions — Implosive Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Extinction Training with LLLT (Experimental): Participants will receive one-session of fear extinction training tailored to the participant's specific fear domain. 15 minutes after fear extinction, participants will receive 8 minutes of Low-Level Laser Therapy stimulation. The laser will be directed at two areas on the forehead: bilateral frontal points Fp1 and Fp2 (on the EEG electrode placement system; to stimulate the vmPFC). Each area will be stimulated for 4 minutes. Treatment will consist of alternating between each of these points after each minute.
  Interventions: Behavioral: Extinction Training; Device: Low-Level Laser Therapy
- Extinction Training with Sham LLLT (Active Comparator): Participants will receive one-session of fear extinction training tailored to the participant's specific fear. 15 minutes after fear extinction, participants will receive 8 minutes of Sham Low-Level Laser Therapy stimulation. The laser will be directed at two areas on the forehead: bilateral frontal points Fp1 and Fp2 (on the EEG electrode placement system). The procedure will consist of alternating between each of these points after each minute. However, each point will receive only a brief (5-second) treatment to the intended site on the forehead, followed by 55 seconds of no treatment, for each one-minute cycle, functioning as a placebo dose of the treatment.
  Interventions: Behavioral: Extinction Training; Device: Sham Low-Level Laser Therapy
- LLLT alone (Experimental): Participants will receive 8 minutes of Low-Level Laser Therapy stimulation. The laser will be targeted first at the left forehead point F3 and then at the right forehead point F4 (on the EEG electrode placement system). F3 corresponds with the left dorsolateral prefrontal cortex and F4 corresponds with the right dorsolateral prefrontal cortex. Each area will be stimulated for 4 minutes. Treatment will consist of alternating between each of these points after each minute.
  Interventions: Device: Low-Level Laser Therapy
- Sham LLLT alone (Sham Comparator): Participants will receive 8 minutes of Sham Low-Level Laser Therapy stimulation. The laser will be targeted first at the left forehead point F3 and then at the right forehead point F4 (on the EEG electrode placement system). The procedure will consist of alternating between each of these points after each minute. However, each point will receive only a brief (5-second) treatment to the intended site on the forehead, followed by 55 seconds of no treatment, for each one-minute cycle, functioning as a placebo dose of the treatment.
  Interventions: Device: Sham Low-Level Laser Therapy

INTERVENTIONS:
Behavioral: Extinction Training — Up to 40 min. of self-directed repeated exposure to a fear-provoking situation.
  Other Names: Exposure Therapy
  Arms: Extinction Training with LLLT; Extinction Training with Sham LLLT
Device: Low-Level Laser Therapy — 1064nm light used to modulate a biological function and induce a therapeutic effect.
  Other Names: LLLT
  Arms: Extinction Training with LLLT; LLLT alone
Device: Sham Low-Level Laser Therapy — Placebo dose version of LLLT.
  Other Names: Sham LLLT
  Arms: Extinction Training with Sham LLLT; Sham LLLT alone

SUMMARY:
There are two specific aims for this study. Aim 1 is to test whether low-level laser therapy (LLLT) can enhance the efficacy of fear extinction training in the modification of pathological fear. Aim 2 is to investigate the efficacy of low-level laser therapy (LLLT) as a stand-alone intervention for anxiety/phobias.

DETAILED DESCRIPTION:
Preliminary research with non-human animals suggests that LLLT (i.e., ultra low doses of transcranial infrared light) can enhance the retention of fear extinction learning by up regulating neuronal metabolic activity when applied to the ventromedial prefrontal cortex (vmPFC). Furthermore, evidence from a previous uncontrolled trial with humans suggests that LLLT (outside the context of extinction training) can lead to a significant decrease in symptoms of depression and anxiety when applied to the right and left dorsolateral prefrontal cortices (dlPFC). The first aim of this study is to test whether LLLT can boost fear reduction after extinction training in humans. A second aim of this study is to investigate the efficacy of LLLT as a stand-alone anxiolytic intervention in a randomized controlled trial.

Individuals between the ages of 18-65 with elevated fear in any of one of four domains (e.g., fear of enclosed spaces, fear of contamination, fear of public speaking, or anxiety sensitivity) are randomly assigned to one of four treatment arms (1) Extinction Training with LLLT, (2) Extinction Training with Sham LLLT, (3) LLLT alone, or (4) Sham LLLT alone.

To determine eligibility, all participants undergo an online prescreen and a face-to-face screening assessment. Participants who qualify for the study then complete a baseline (pre-treatment) assessment, followed immediately by the treatment procedure and a post-treatment assessment. Participants return to the lab an average of 14 days after treatment to complete a follow-up assessment. Participants complete two behavioral approach tests (in the treatment context and in the generalization context) at baseline, post-treatment, and follow-up, and a battery of self-report questionnaires at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65
2. Behavioral Approach Test (BAT) peak fear rating equal to or greater than 50/100 on both BATs (i.e., treatment and generalization contexts).

Exclusion Criteria:

1. High risk for suicide as determined by a clinical assessment, which will occur if a participant indicates that they are currently experiencing suicidal ideation on the depression module of the Mini International Neuropsychiatric Inventory, or on item 9 of the Beck Depression Inventory.
2. Psychotropic medication taken within the past 4 weeks.
3. Currently Receiving treatment for the fear domain in question.
4. Presence of a medical condition (i.e., pregnancy, seizure disorder, respiratory disorder, cardiovascular disease) that would contraindicate participation in one or more treatment or assessment activities as determined by a Medical History Questionnaire.
5. Active neurological condition (such as epilepsy or stroke) as determined by a Medical History Questionnaire.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Behavioral Approach Test- Generalization Context | Baseline (Day 1); Post-treatment (Day 1; immediately after treatment); Follow-up (2 weeks, average of 14 days after treatment)
  Change in fear response as indicated by behavioral approach and peak subjective fear ratings (0-100) in a generalization context (different from the treatment context) from baseline to follow-up.

SECONDARY OUTCOMES:
Behavioral Approach Test - Treatment Context | Baseline (Day 1); Post-treatment (Day 1; immediately after treatment); Follow-up (2 weeks, average of 14 days after treatment)
  Change in fear response as indicated by behavioral approach and peak subjective fear ratings (0-100) in a generalization context (different from the treatment context) from baseline to post-treatment.
Beck Depression Inventory-II (BDI-II) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in depression symptoms from baseline to follow-up.
Beck Anxiety Inventory (BAI) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in anxiety symptoms from baseline to follow-up.
Claustrophobia Questionnaire (CLQ) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in claustrophobic cognitions from baseline to follow-up (for participants in the fear of enclosed spaces domain).
Claustrophobia Concerns Questionnaire (CCQ) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in claustrophobic cognitions from baseline to follow-up (for participants in the fear of enclosed spaces domain).
Obsessive Compulsive Inventory-Revised (OCI-R) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in obsessional symptoms from baseline to follow-up (for participants in the fear of contamination domain).
Washing Threat Questionnaire (WTQ) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in threat perceptions related to not being able to wash hands from baseline to follow-up (for participants in the fear of contamination domain).
Liebowitz Social Anxiety Scale Self Report Version (LSAS-SR) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in anxiety and avoidance for social situations from baseline to follow-up (for participants in the fear of public speaking domain).
Speech Anxiety Thoughts Inventory (SATI) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in maladaptive cognitions associated with speech anxiety from baseline to follow-up (for participants in the fear of public speaking domain).
Anxiety sensitivity Index (ASI-3) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in fear ratings of physical, cognitive, and social anxiety reactions or sensations from baseline to follow-up (for participants in the anxiety sensitivity domain).
Body Sensations Questionnaire (BSQ) | Baseline (Day 1; beginning of first visit); Follow-up (2 weeks, average of 14 days after treatment)
  Change in fear ratings in relation to somatic sensations from baseline to follow-up (for participants in the anxiety sensitivity domain).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Telch, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- Laboratory for the Study of Anxiety Disorders, Austin, Texas, United States

REFERENCES:
- [Result] Zaizar ED, Papini S, Gonzalez-Lima F, Telch MJ. Singular and combined effects of transcranial infrared laser stimulation and exposure therapy on pathological fear: a randomized clinical trial. Psychol Med. 2023 Feb;53(3):908-917. doi: 10.1017/S0033291721002270. Epub 2021 Jul 21. PMID 34284836
- See also: Primary Outcomes Results Paper — https://doi.org/10.1017/S0033291721002270